CLINICAL TRIAL: NCT05205629
Title: A Real-world Clinical Study of Donafenib Combined With TACE as a Basis for the Treatment of Unresectable Hepatocellular Carcinoma
Brief Title: A Real-world Study of Donafenib Combined With TACE-based Treatment in Patients With Unresectable HCC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: B2021-640R
Record Dates: First submitted 2021-12-23; First posted 2022-01-25 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-01

CONDITIONS: Hepatocellular Carcinoma; Donafenib
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — donafenib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Donafenib + TACE
  Interventions: Drug: Donafenib combined with TACE

INTERVENTIONS:
Drug: Donafenib combined with TACE — Donafenib(200mg bid po) combined with TACE
  Other Names: Donafenib plus TACE

SUMMARY:
This study is a prospective, single-center, observational real-world study. It is planned to enroll 150 patients with unresectable hepatocellular carcinoma treated with Donafenib combined with TACE-based treatment, so as to observe and evaluate the efficacy and safety of Donafenib combined with TACE-based treatment in patients with unresectable HCC.

ELIGIBILITY:
Inclusion Criteria:

1. Patients voluntarily entered the study and signed informed consent form (ICF);
2. Age: Be at least 18 years old and and there is no limit on the gender;
3. Clinically or histologically diagnosed as unresectable HCC;
4. There is at least one measurable lesions that meet the mRECIST standard;
5. Child-pugh classification A or B (score≤7);
6. The maximum number of TACE procedures allowed before enrolment was 2. All of those patients who had a history of prior TACE achieved complete response by previous TACE, but recurred more than 6 months later at the study entry
7. ECOG : 0 ~ 2 ;
8. Before the patients were enrolled in the study, doctors had decided to treat them with donafenib in combination with TACE.

Exclusion Criteria:

1. Donafenib forbidden population:

   * Those who are allergic to any component of the medicine;
   * Active bleeding;
   * Active peptic ulcer;
   * Hypertension not controlled by drugs;
   * Those with severe liver insufficiency.
2. Medical conditions that affect absorption, distribution, metabolism, or clearance of the study drug (e.g., severe vomiting, chronic diarrhea, intestinal obstruction, absorption disorders, etc.);
3. Patients with a clear past history of neurological or psychiatric disorders;
4. The patient had been treated with another study drug or study device in the 4 weeks prior to initial dosing;
5. Pregnant or breastfeeding women, and women or men with fertility who are unwilling or unable to take effective contraceptive measures;
6. Unable to follow the research protocol for treatment or scheduled follow-up;
7. Any other researcher who thinks they cannot be included.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Source of subjects: Unresectable HCC patients treated with Donafenib and TACE from Zhongshan Hospital Affiliated to Fudan University.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-01-30 (Actual); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | an expected average of 8 months
  Defined as the time from the start of enrollment to the occurrence of disease progression that cannot be treated by TACE or death due to various reasons.

SECONDARY OUTCOMES:
Objective response rate | an expected average of 12 months
  evaluated by investigators with mRECIST
Disease control rate | an expected average of 12 months
  evaluated by investigators with mRECIST
Time to untreatable progression | an expected average of 12 months
  It is defined as the time when a tumor that cannot be treated by TACE progresses, deteriorates to Child-pugh C, or appears extrahepatic metastasis.
Overall survival | an expected average of 18 months
  The time from enrollment to the death from any cause
The incidence of AEs and SAEs by NCI-CTCAE v5.0 | an expected average of 18 months
  Safety index
Conversion rate | an expected average of 18 months
  Defined as the proportion of patients who can undergo radical surgical resection through conversion therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University, Shanghai, China